CLINICAL TRIAL: NCT03398161
Title: Ultra Low Dose Radiation for Local Treatment of Cutaneous Mycosis Fungoides
Brief Title: Ultra Low Dose Radiation Therapy in Treating Patients With Mycosis Fungoides
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0276; NCI-2018-00861 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0276 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Localized Skin Lesion; Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (ultra low dose radiation therapy) (Experimental): Patients undergo ultra low dose radiation therapy at the discretion of the treating physician.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo ultra low dose radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well ultra low dose radiation therapy works in treating patients with mycosis fungoides. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving ultra low doses of radiation may help control the disease and reduce side effects compared to treatment with higher doses.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of low dose radiation in the management of cutaneous mycosis fungoides (MF), measured as any local control for each lesion at 12 (+/- 2) weeks after the treatment, in patients with stage IA - IVB cutaneous MF.

SECONDARY OBJECTIVES:

I. To evaluate complete response (CR) rates at 12 (+2) weeks and beyond.

II. To evaluate the persistence of response (CR, partial response [PR], stable disease, or progressive disease) in the treated lesion beyond 12 (+2) weeks.

III. To evaluate overall survival.

IV. To evaluate progression free survival.

V. To evaluate patient symptom relief.

VI. To evaluate the toxicity of radiation to the skin.

VII. To assess if number of previous therapies including chemotherapy, targeted therapy, topical therapy, or total skin radiation affects the response.

VIII. To characterize the microbiome of mycosis fungoides patient within both the lesion and unaffected skin.

IX. To characterize shifts in the microbiome that occur after radiation therapy.

OUTLINE:

Patients undergo ultra low dose radiation therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 4-6 and 10-14 weeks, every 3 months for 6-8 months, then every 6-12 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed MF with cutaneous involvement.

  * Patients must have clinically measurable disease of at least 1 lesion on physical (skin) exam.
  * If a patient has a prior pathological diagnosis of MF and is clinically diagnosed with a new lesion, the new lesion is eligible for enrollment without additionally biopsy confirmation.
* Lesions of any surface span as long as =< 1 cm in maximal height measured from the skin surface for which local control is desired are eligible; a single patient may have multiple eligible lesions that are individually enrolled for the study.
* All stages of disease (IA through IVB) where radiation therapy is being considered for local control are eligible. Patients who are concomitantly undergoing systemic therapy for more advanced stage disease are eligible.
* Patients who are concomitantly undergoing systemic therapy for more advanced stage disease are eligible.
* Female patients of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [hCG]) within 2 weeks of protocol entry if the patient is unsure of their pregnancy status. Patient signature declaring that they are not pregnant on the informed consent for treatment that is used in the Department of Radiation Oncology is also an acceptable substitution for a serum pregnancy test.
* Patients who are receiving or are planned to start topical chemotherapeutics, retinoids or imiquimod to other lesions that are not planned for enrollment are eligible; however, the lesion being considered for enrollment should not be under active therapy with these topical agents immediately prior to enrollment.

  * Use of topical chemotherapeutics, retinoids or imiquimod on the lesion that is a candidate for enrollment must be halted at least 24 hours prior to enrollment in the study.

Exclusion Criteria:

* Pregnant patients do not meet inclusion criteria for radiation therapy.

  * Patients who subsequently become pregnant may continue follow up within the protocol, but a negative urine pregnancy test will need to be obtained before additional lesions may be enrolled.
* Patients with active lupus or scleroderma
* Lesions with a height > 1 cm measured from the skin surface are not eligible for this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Local cutaneous control | At 12 (+/-2) weeks after initial treatment
  Defined as local control of the treated lesion within the radiation treatment field, which will be categorized as either complete response or partial response of the lesion within the radiation treatment field. The control rate will be estimated along with 95% confidence intervals. The association between control rate and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate. For each patient, the number of lesions under control will be summarized individually. Since there may be multiple lesions per patient, a generalized linear mixed model will be utilized to assess the clinical factor effect (e.g. previous therapies) on control rate after considering the dependence among the lesions within each patient.

SECONDARY OUTCOMES:
Stable disease, progressive disease, or local regional control (local control within the radiation field margin but not encompassing the original treated lesion) | Up to 2 years
  Will be described with frequency tables.
Overall survival | From initiation of treatment until death, assessed up to 2 years
  Will be described with frequency tables. Will be conducted using the Kaplan Meier Method.
Progression free survival | From treatment until progression or death, assessed up to 2 years
  Will be described with frequency tables. Will be conducted using the Kaplan Meier Method.
Frequency/severity of skin toxicity | Up to 14 weeks
  Defined by patient reported symptom surveys. Toxicity type (acute or chronic), severity and attribution will be summarized for each patient using frequency tables. Different time points (e.g. pre and post-treatment) will be compared using a paired t-test or Wilcoxon signed rank test as appropriate.
Microbiome analysis | Up to 2 years
  Will be described with frequency tables.
Quality of life | Up to 2 years
  Will be assessed by the Skindex-16 survey. Will be summarized by domains. Different time points (e.g. pre and post-treatment) will be compared using a paired t-test or Wilcoxon signed rank test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina S Dabaja, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org